CLINICAL TRIAL: NCT06025370
Title: Measurement of Pressures Generated During Different Prone Positions in Healthy Volunteers
Brief Title: Pressures During Prone Positions in Healthy Volunteers
Acronym: HEALTHY-PRONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CHRO-2022-13
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Pressure Ulcer
Keywords: Healthy Volunteer; Pressure Mapping; ARDS; Prone Position
MeSH Terms: conditions — Pressure Ulcer | interventions — Prone Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swimmer Position (Experimental)
  Interventions: Other: Prone Position
- Arms at side (Active Comparator)
  Interventions: Other: Prone Position

INTERVENTIONS:
Other: Prone Position — All healthy volunteers will be positioned in prone position, on a bed equipped with a mapping pressure system.
  The volunteers will spend 5 minutes in each of the positions corresponding to the study groups.

SUMMARY:
Prone positioning (PP) reduces mortality in the most severe cases of acute respiratory distress syndrome (ARDS). Despite the benefits of PP, this technique presents adverse effects such as an increased risk of bedsores, linked to the duration, which must be around 16 consecutive hours.

There are 2 PP techniques:

1. Positioning with arms alongside the body
2. Swimmer's position At present, no study compares or has compared prospectively, the impact of the type of position used during ventral decubitus on mortality and the incidence of pressure sores, nor on secondary effects in intensive care.

Pressure transducers are available for instantaneous measurement of pressures between 2 interfaces. The investigators have acquired a pressure-measuring device, a mattress topper which is attached to the resuscitation mattress and which, connected to a PC, provides a live display of the pressures between the patient and the mattress.

The investigators would like to use their device to measure pressures during these 2 PP in healthy volunteers, which would enable them to obtain the world's first data on the real pressures generated during PP.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Major volunteer

Exclusion Criteria:

* Volunteers with cervical mobility problems preventing them from rotating their head 90°
* Volunteers with scapulohumeral joint mobility problems preventing them from performing 90° elevation/abduction.
* Pregnant volunteer (confirmed by a blood sample test or a positive pregnancy test).
* Volunteer not affiliated to a French social security system
* Volunteer protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Skin/Bed pressures | 5 minutes
  Obtain pressure values for both prone position techniques on pressure sore risk zones (face/shoulders/hips/knees/feet)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume FOSSAT, Msc, Principal Investigator — CHU ORLEANS
Locations (1):
- Centre Hospitalier Régional d'Orléans, Orléans, Centre-Val de Loire, France

IPD SHARING:
Plan to Share IPD: No